CLINICAL TRIAL: NCT06646003
Title: Reference Values and Determinants of 6-minute Walk Test Distance in Turkish Patients With Chronic Stroke: A Multicenter Cross-sectional Study
Brief Title: Reference Values and Determinants of 6-minute Walk Test
Status: Completed | Type: Observational
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Merve Örücü Atar, Associate professor, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Other Study IDs: 1-24-599
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2024-11

CONDITIONS: Stroke
Keywords: walking
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- stroke group: patients with chronic stroke
  Interventions: Other: Evaluation of 6-minute walking distance and related factors in patients with chronic stroke

INTERVENTIONS:
Other: Evaluation of 6-minute walking distance and related factors in patients with chronic stroke — Evaluation of 6-minute walking distance and related factors in patients with chronic stroke.

SUMMARY:
The first aim of this study was to investigate the reference values of 6-minute walk test (6MWT) distance in patients with chronic stroke. The second aim was to determine the factors predicting 6MWT distance in patients with chronic stroke.

DETAILED DESCRIPTION:
There may be large variations in the distance of 6MWT according to the stroke severity. Investigation of factors related to 6MWT may be helpful in determining and targeting appropriate strategies for gait rehabilitation. Accordingly, the first aim of this study was to investigate the reference values of 6-minute walk test (6MWT) distance in patients with chronic stroke. The second aim was to determine the factors predicting 6MWT distance in patients with chronic stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Having first ever stroke
2. The time elapsed after the stroke is more than 6 months and less than 10 years
3. 18-80 years old
4. Those who could walk independently with no assistance or device and who could walk with an intermittent or continuous light touch to assist balance or coordination

Exclusion Criteria:

Exclusion Criteria:

1. A history of severe musculoskeletal, cardiopulmonary, or psychiatric disease that can inhibit measurements
2. Patients who had received a neurologic diagnosis other than stroke, such as Parkinson's disease or multiple sclerosis
3. Patients with impaired level of consciousness and evidence of gross cognitive impairment (Scored below 10 points in the Mini-Mental State Examination

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with chronic stroke
Sampling Method: Non-Probability Sample
Enrollment: 341 (Actual)
Dates: Start 2024-11-30 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2025-11-25 (Actual)

PRIMARY OUTCOMES:
6-minute walk test (6MWT) | through study completion, an average of one month
  6MWT will be used to evaluate the walking endurance. A 30-m indoor walkway will be used to conduct the test. The maximal distance covered at the end of the 6MWT will be recorded.

SECONDARY OUTCOMES:
Functional ambulation scale (FAC) | through study completion, an average of one month
  Patients will be classified by walking ability using FAC has six levels (0 to 5) that are classified according to the walking ability on the basis of the amount of physical support required, which are as follows: nonfunctional ambulatory(FAC 0); ambulatory, continuous manual contact to support body weight as well as to maintain balance or to assist coordination (FAC 1); ambulatory [level I], intermittent or continuous light touch to assist balance or coordination (FAC 2); ambulatory, dependent on supervision (FAC 3); ambulatory, independent, level surface only (FAC 4); and ambulatory, independent (FAC 5).
Brunnstrom motor recovery staging | through study completion, an average of one month
  Upper extremity, hand and lower extremity motor recovery will be assessed using the Brunnstrom 6 sequential stages of motor recovery.
Modified Ashworth Scale (MAS) | through study completion, an average of one month
  The Modified Ashworth Scale will be used to measure the severity of knee extensor, knee flexor and ankle plantar flexor spasticity. MAS scores will be added together to give a total MAS score. MAS is graded from 0 to 4. A score of 0 indicates no increase at all in muscle tone, and 4 indicates that the joint is rigid in flexion or extension.
Beck depression inventory (BDI) | through study completion, an average of one month
  The beck depression inventory (BDI) will be used to evaluate depression. The BDI consists of 21 questions about how the subject has been feeling in the last week. Each question has a set of at least four possible answers, ranging in intensity. A value of 0-3 is assigned for each answer, and the total score is compared with a key to determine the severity of depression .The standard cut off values are as follows: 0-9, minimal depression; 10-18, mild depression; 19-29, moderate depression; and 30-63, severe depression.
Mini-mental state examination (MMSE) | through study completion, an average of one month
  The mini-mental state examination will be used to describe mental and cognitive functions.
Star cancellation test | through study completion, an average of one month
  Star cancellation test will be used to describe neglect phenomenon.
Barthel Index | through study completion, an average of one month
  Activities of daily living (ADL) will be assessed using the Barthel Index. The Barthel Index consists of 10 items that measure a person's daily functioning, specifically ADL and mobility. The items include feeding, bathing, grooming, dressing, toileting, transferring, walking on a level surface, going up and down stairs, and continence of bowel and bladder. A patient with a maximum score of 100 points is defined as continent, able to eat and dress independently, able to walk at least a block, and able to go up and down stairs.
Berg Balance Scale (BBS) | through study completion, an average of one month
  Balance ability will be tested using the Berg Balance Scale (BBS), which includes 14 functional balance items, with scores ranging from 0 to 56 points; better balance is indicated by a higher score.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Gaziler Physical Medicine and Rehabilitation Education and Research Hospital, Ankara, Turkey (Türkiye)